CLINICAL TRIAL: NCT05259007
Title: The Effect of Propolis and Nutritional Education in Patients With H. Pylori on Gastrointestinal Symptoms
Brief Title: Effect of Propolis on Patients Infected With H. Pylori
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fatma Zehra Arvas (Other)
Collaborators: Apipark Beekeeping (Unknown)
Responsible Party: Sponsor-Investigator, Fatma Zehra Arvas, dietitian, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: E-77979112-424.04.01-82
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: H.Pylori,Propolis,Nutritional Education,PUD
MeSH Terms: interventions — Sodium Chloride; Lactic Acid

STUDY DESIGN:
Intervention Model Description: 96 patients divided into three groups: Group 1 propolis with lactic acid extract on top of the treatment given by doctor Group 2 Lactic acid extract on top of the treatment by the doctor Group 3 the treatment given by the doctor and placebo treatment
Who Masked: Participant, Investigator
Masking Description: Double blind randomized controlled trial study will be utilized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group 1 propolis with lactic acid extract on top of the treatment given by doctor
  Interventions: Dietary Supplement: propolis solved in lactic acid solvent; Drug: Amoxicillin-Clarithromycin-Lansoprazole
- Group 2 (Other): Grorup 2 Lactic acid extract on top of the treatment by the doctor
  Interventions: Drug: Amoxicillin-Clarithromycin-Lansoprazole; Other: Lactic acid
- Group 3 (Placebo Comparator): Group 3 the treatment given by the doctor and placebo treatment
  Interventions: Drug: Amoxicillin-Clarithromycin-Lansoprazole; Other: IV saline 0.9%

INTERVENTIONS:
Dietary Supplement: propolis solved in lactic acid solvent — propolis given as a dietary supplement which was solved in a lactic acid solvent.
  Arms: Group 1
Drug: Amoxicillin-Clarithromycin-Lansoprazole — H pylori eradication treatment
Other: IV saline 0.9% — Physiological serum solution is given as a placebo
  Arms: Group 3
Other: Lactic acid — given to determine if the improvement of the symptoms are due to propolis or the solvent
  Arms: Group 2

SUMMARY:
This research aims to contribute to the literature by researching the effect of propolis as an add-on treatment and nutritional education on patients with H pylori and the alleviation of gastrointestinal symptoms.In order to achieve this, we offered propolis and educational nutrion programme to our 96 patients and check on their symptoms on a regular basis to note any improvement by measuring the alleviation using GSRS.

DETAILED DESCRIPTION:
The informed voluntary consent was taken from the patients who agreed to attend the research and the patients, Group 1 propolis with lactic acid extract on top of the treatment given by doctor Group 2 Lactic acid extract on top of the treatment by the doctor Group 3 the treatment given by the doctor and placebo treatment ,will be distributed by the method of randomized double blind trial.The patients will be provided with 500 mg (≌60 drops/day) of propolis or propolis with lactic acid extract in the morning,afternoon and evening for 14 days.The face-to-face Survey data collection method will be utilized and the researcher inform the patients about the diet and nutrition education against pylori and propolis.The presentation for the Patient Education and Propolis is given in the appendix.

The survey form consists of 4 parts; descriptive general information,eating habits,Gastrointestinal Symptoms Rating Scale (GSRS) and the frequency of The consumption of particular food. In order to rate the gastrointestinal symptoms of the patients the GSRS scale which was validated and deemed reliable in Turkish will be used The foods that increase the frequency of gastrointestinal symptoms such as spicy foods,chocolate,Chips,carbonated drinks,citrus fruits are also questioned in terms of frequency of consumption.

In order to investigate the patients adherence to the study, reminders will be taking place by giving them a call two times a week. At the end of the intervention period,GSRS scale will be reused to assess the patients.

ELIGIBILITY:
Inclusion Criteria:

* The detection of H pylori infection by a specialized physician.

Exclusion Criteria:Bees and bees products allergies and the patients who use drugs that has bleomycin as an active compound will be excluded as it was found in the rats that these types of antitumor drugs can interact with propolis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-02-22 (Estimated); Primary Completion 2022-03-23 (Estimated); Study Completion 2022-04-05 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale | 14 days
  The follow up of the patients are done by Gastrointestinal Symptom Rating Scale

IPD SHARING:
Plan to Share IPD: No
It was decided that only the investigators could access the participants data and it will remain confidential to all other outsiders.

REFERENCES:
- See also: Propolis polyphenolic compounds affect the viability and structure of Helicobacter pylori in vitro — https://www.scielo.br/j/rbfar/a/3LHfSb5j7gcxJNPTFTq6ZLK/abstract/?lang=en
- See also: CHARACTERIZATION OF Helicobacter pylori, RESEARCH OF INHIBITION EFFECTS OF HONEY AND PROPOLIS SAMPLES ON BACTERIA AND UREASE — http://acikerisim.erdogan.edu.tr/xmlui/handle/11436/133
- See also: Reliability and Validity of the Turkish Version of the Gastrointestinal Symptom Rating Scale — https://journals.lww.com/gastroenterologynursing/Fulltext/2017/01000/Reliability_and_Validity_of_the_Turkish_Version_of.6.aspx?casa_token=2oaHZJdvgH8AAAAA:rsEjdqS5cHOruhlESJivfm2cklYtHUgZBVvklYF_amoNHqZ-xP8OeZexcvYZVszCCfFMxF5-bEcN51yvm3o_6Q1btg
- See also: The Effect of Propolis as a Functional Product on Health — https://dergipark.org.tr/en/download/article-file/1205293